CLINICAL TRIAL: NCT03774771
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, 6-week Dose-Ranging Study to Assess the Safety, Pharmacokinetics, and Clinical Effects of an Oral Calcimimetic Agent (AMG 073) in Primary Hyperparathyroidism
Brief Title: Safety, Pharmacokinetics, and Clinical Effects of Cinacalcet (AMG 073) in Primary Hyperparathyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 00980125
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): In Part 1 participants received placebo capsules orally once a day for 6 weeks. In Part 2 participants received placebo capsules twice a day for 15 days.
  Interventions: Drug: Placebo
- Cinacalcet 50 mg QD (Experimental): In Part 1 participants received 50 mg cinacalcet capsules orally once a day (QD) for 6 weeks. In Part 2 participants received 30 mg cinacalcet capsules twice a day for 15 days.
  Interventions: Drug: Cinacalcet
- Cinacalcet 75 mg QD (Experimental): In Part 1 participants received 75 mg cinacalcet capsules orally once a day (QD) for 6 weeks. In Part 2 participants received 40 mg cinacalcet capsules twice a day for 15 days.
  Interventions: Drug: Cinacalcet
- Cinacelcet 100 mg QD (Experimental): In Part 1 participants received 100 mg cinacalcet capsules orally once a day (QD) for 6 weeks. In Part 2 participants received 50 mg cinacalcet capsules twice a day for 15 days.
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: Cinacalcet — Capsule for oral administration
  Other Names: AMG 073; Sensipar®; Mimpara®
  Arms: Cinacalcet 50 mg QD; Cinacalcet 75 mg QD; Cinacelcet 100 mg QD
Drug: Placebo — Capsules for oral administration
  Arms: Placebo

SUMMARY:
The primary objective was to assess the safety and tolerability of cinacalcet in adults with primary hyperparathyroidism (HPT) when administered as a single oral once daily doses for 6 consecutive weeks and twice daily for 15 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age at screening. In Part 1, females must be postmenopausal (at least 12 months since last menstrual period) or surgically sterile.

   In Part 2, all qualified females replacing a Part 1 subject (i.e., naïve subjects), regardless of reproductive status, may participate if, in the opinion of the principal investigator, an appropriate effective contraceptive method is used throughout the study. All females must have a negative serum pregnancy test within 28 days prior to Baseline (Parts 1 and 2).
2. Men and women participating in this study must agree to use, in the opinion of the principal investigator, highly effective contraceptive measures throughout the study. All females who are pregnant or breast-feeding are excluded. All subjects must notify the principal investigator if they or their partner suspects a pregnancy.
3. Diagnosis of primary HPT. A plasma intact PTH concentration ≥ 45 pg/mL on at least two occasions at least 1 week apart during the 12 months prior to baseline (at least one of these determinations should be made during screening), and a corrected total serum calcium concentration (for each 1 g/dL decrease in albumin level below 4.0 g/dL, the calcium value should be increased by 0.8 mg/dL) greater than the upper limit of normal, but no greater than 12.5 mg/dL.
4. Acceptable renal function, with an estimated creatinine clearance > 50 ml/min as determined by the Cockroft and Gault equation.
5. Acceptable hepatic function, defined as serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin < 2 times the upper limit of normal.
6. Fasting (8 hours) serum glucose ≤ 130 mg/dL and hemoglobin Alc within the central laboratory's normal range.
7. Hematology panel, serum clinical chemistry and urinalysis results within normal ranges
8. Chest x-ray without evidence of active, infectious, inflammatory or malignant process.

Exclusion Criteria:

1. Any unstable medical condition, defined as having been hospitalized within 28 at prior to baseline, or otherwise unstable in the judgement of the investigator.
2. Received within 21 day prior to baseline, therapy with systemic glucocorticoids, lithium, tricyclic antidepressants, thioridazine, haloperidol, flecainide, or other drugs with a narrow therapeutic index that are primarily metabolized by hepatic cytochrome P450 CYP 2D6, drugs that affect renal tubular calcium handling (e.g. thiazide or loop diuretics), and drugs that affect bone metabolism (e.g. calcitonin, selective estrogen receptor modulators [SERMs])
3. Received, within 90 days prior to Baseline, chronic therapy with bisphosphonates or fluoride.
4. Known alcohol abuse, or use of illicit drugs, within 12 months prior to Baseline
5. Experienced a myocardial infarction (MI) within 6 months prior to Baseline
6. A ventricular rhythm disturbance requiring current treatment
7. Received investigational drugs within 28 days prior to Baseline
8. A history of seizures within 12 months prior to Baseline
9. A history (within 5 years) of malignancy of any type, other than nonmelanomatous skin cancers or in situ cervical cancer
10. A gastrointestinal disorder that may be associated with impaired absorption of orally administered medications
11. A Body Mass Index (BMI) < 15 or > 40, obtained during screening
12. An inability to swallow capsules
13. Sarcoidosis, tuberculosis, or other diseases known to cause hypercalcemia
14. Fasting spot urine calcium/creatinine ratio (mg) < 0.05
15. A psychiatric disorder that would interfere with understanding and giving informed consent or compliance with protocol requirements
16. Any other condition that might reduce the chance of obtaining data (eg, known poor compliance) required by the protocol or that might compromise the ability to give truly informed consent.
17. For Part 2, a subject from Part 1 who discontinued treatment early

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 1998-09-29 (Actual); Primary Completion 1999-12-13 (Actual); Study Completion 1999-12-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events in Part 1 and Part 2 | 6 weeks in Part 1 and 15 days in Part 2

SECONDARY OUTCOMES:
Percent Change from Baseline in Serum Calcium Concentration | Baseline and days 8, 15, 16, 29, 43, and 50 in Part 1 and days 1, 8, 15, and 22 in Part 2.
Area Under the Serum Calcium Concentration-time Curve from 0 to 24 Hours After Dosing (AUC0-24) in Part 1 | Days 1, 8, and 43: Predose, 1, 2, 4, 8, 12, and 24 hours post dose
Area Under the Serum Calcium Concentration-time Curve from 0 to 12 Hours After Dosing (AUC0-12) in Part 2 | Days 1 and 15: Predose, 1, 2, 4, 8, 12, 13, 14, 16, 20, and 24 hours postdose
Minimum Serum Calcium Concentration in Part 1 | Days 1, 8, and 43: Predose, 1, 2, 4, 8, 12, and 24 hours postdose
Minimum Serum Calcium Concentration in Part 2 | Days 1 and 15: Predose, 1, 2, 4, 8, 12, 13, 14, 16, 20, and 24 hours postdose
Cumulative Time When Serum Calcium was Below Baseline During the 24-hour Dosing Interval in Part 1 | Days 1, 8, and 43: Predose, 1, 2, 4, 8, 12, and 24 hours post dose
Cumulative Time When Serum Calcium was Below Baseline During the 12-hour Dosing Interval in Part 2 | Days 1 and 15: Predose, 1, 2, 4, 8, 12, 13, 14, 16, 20, and 24 hours postdose
Cumulative Time Over the Day When Serum Calcium was ≤ 10.3 mg/dL In Part 1 | Days 1, 8, and 43: Predose, 1, 2, 4, 8, 12, and 24 hours post dose
Cumulative Time Over the Day When Serum Calcium was ≤ 10.3 mg/dL In Part 2 | Days 1 and 15: Predose, 1, 2, 4, 8, 12, 13, 14, 16, 20, and 24 hours postdose
Percent Change from Baseline in Plasma Intact parathyroid Hormone (iPTH) Concentration | Baseline and days 8, 15, 16, 29, 43, and 50 in Part 1 and days 1, 8, 15, and 22 in Part 2.
Area Under the Plasma iPTH Concentration-time Curve from 0 to 24 Hours After Dosing (AUC0-24) in Part 1 | Days 1, 8, and 43: Predose, 1, 2, 4, 8, 12, and 24 hours post dose
Area Under the Plasma iPTH Concentration-time Curve from 0 to 12 Hours After Dosing (AUC0-12) in Part 2 | Days 1 and 15: Predose, 1, 2, 4, 8, 12, 13, 14, 16, 20, and 24 hours postdose
Minimum iPTH Concentration in Part 1 | Days 1, 8, and 43: Predose, 1, 2, 4, 8, 12, and 24 hours postdose
Minimum iPTH Concentration in Part 2 | Days 1 and 15: Predose, 1, 2, 4, 8, 12, 13, 14, 16, 20, and 24 hours postdose
Time of Minimum iPTH Concentration in Part 1 | Days 1, 8, and 43: Predose, 1, 2, 4, 8, 12, and 24 hours postdose
Time of Minimum iPTH Concentration in Part 2 | Days 1 and 15: Predose, 1, 2, 4, 8, 12, 13, 14, 16, 20, and 24 hours postdose
Cumulative Time When iPTH was Below Baseline During the 24-hour Dosing Interval in Part 1 | Days 1, 8, and 43: Predose, 1, 2, 4, 8, 12, and 24 hours post dose
Cumulative Time When iPTH was Below Baseline During the 12-hour Dosing Interval in Part 2 | Days 1 and 15: Predose, 1, 2, 4, 8, 12, 13, 14, 16, 20, and 24 hours postdose
Cumulative Time iPTH was Below 45 pg/mL in Part 1 | Days 1, 8, and 43: Predose, 1, 2, 4, 8, 12, and 24 hours post dose
Cumulative Time iPTH was Below 45 pg/mL in Part 2 | Days 1 and 15: Predose, 1, 2, 4, 8, 12, 13, 14, 16, 20, and 24 hours postdose
Percent Change from Baseline in Serum Calcitonin Concentration | Baseline and days 8, 15, and 43 in Part 1
Percentage of Participants with Serum Calcitonin Concentration Less than 10 pg/mL | Baseline and days 8, 15 and 43 in Part 1
Percent Change from Baseline in Bone-specific Alkaline Phosphatase (BALP) Concentration | Baseline and days 15 and 43 in Part 1 and days 1, 8, and 15 in Part 2
Percentage of Participants with BALP Concentration Within Normal Range | Baseline and days 15 and 43 in Part 1 and days 1, 8, and 15 in Part 2
  Normal range of BALP is 2.9 to 20.1 ng/mL for men 20 to 79 years of age and and 3.7 to 20.9 ng/mL for women 20 to 79 years of age.
Percent Change from Baseline in Serum N-telopeptide (NTx) Concentration | Baseline and days 8 and 15 in Part 1
Percentage of Participants with Serum NTx Concentration Within Normal Range | Baseline and days 8 and 15 in Part 1
  Normal range of serum NTx is 5.4 to 24.2 nmoL bone collagen equivalents (BCE)/L for men, 6.2 to 19.0 nmoL BCE/L for premenopausal women, and 5.3 to 35.8 nmol BCE/L for postmenopausal women (≥ 55 years).
Percent Change from Baseline in Urinary NTx Concentration | Baseline and days 15 and 43 in Part 1 and days 1, 8, and 15 in Part 2
Percentage of Participants with Urinary NTx Concentration Within Normal Range | Baseline and days 15 and 43 in Part 1 and days 1, 8, and 15 in Part 2
  Normal range of urinary NTx is is 0.0 to 85.0 nmoL BCE/mmoL creatinine for men, 5.0 to 65.0 nmoL BCE/mmoL creatinine for premenopausal women, and 0.0 to 130.0 nmoL BCE/mmoL creatinine for postmenopausal women [≥ 55 years).
Percent Change from Baseline in Urinary Calcium/Creatinine Ratio | Baseline and days 8 and 15 in Part 1
Percent Change from Baseline in Urinary Calcium Concentration | Baseline and days 15 and 43 in Part 1 and days 1, 8, and 15 in Part 2
Percentage of Participants with Urinary Calcium Concentration Within Normal Range | Baseline and days 15 and 43 in Part 1 and days 1, 8, and 15 in Part 2
  Normal range of urinary calcium is 50 to 300 mg/24 hours.
Percent Change from Baseline in 1,25-Dihydroxy Vitamin D | Baseline and days 8 and 43 in Part 1 and days 1 and 15 in part 2
Percentage of Participants with 1,25-Dihydroxy Vitamin D Concentration in the Normal Range | Baseline and days 8 and 43 in Part 1 and days 1 and 15 in part 2
  The normal range for 1,25-dihydroxy vitamin D3 is 16.0 to 65.0 pg/mL.
Percent Change from Baseline in Urinary and Serum Phosphorus Concentrations | Baseline and days 8, 15, and 22 in Part 2